CLINICAL TRIAL: NCT01271179
Title: Study of Sequential Perfusion of Liver Grafts With Low-viscosity and High-viscosity Preservation Solutions to Decrease the Incidence of Nonanastomotic Biliary Strictures After Liver Transplantation
Brief Title: Study of Sequential Perfusion of Liver Grafts to Prevent Nonanastomotic Biliary Strictures After Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Zhi-Hai Peng/ vice-president of Shanghai First People's Hospital, Shanghai First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SFPH04618
Record Dates: First submitted 2010-12-30; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2010-12

CONDITIONS: Liver Transplantation; Transplant Recipient
Keywords: orthotopic liver transplantation; preservation solution; peribiliary plexus; nonanastomotic biliary strictures; primary non-function
MeSH Terms: interventions — University of Wisconsin-lactobionate solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sequential perfusion (Active Comparator): sequential perfusion of liver grafts with low-viscosity improved Ross solution and high-viscosity UW solution.
  Interventions: Procedure: sequential perfusion with ipv Ross solution and UW solution
- sole perfusion (Placebo Comparator): sole perfusion of liver grafts with high-viscosity UW solution only
  Interventions: Procedure: sole perfusion with UW solution

INTERVENTIONS:
Procedure: sequential perfusion with ipv Ross solution and UW solution — Totally 6 L of ipv Ross solution were initially infused (aortic: portal=1:1), followed by 2 L of cold UW solution infusion (aortic: portal=1:1).
  Arms: sequential perfusion
Procedure: sole perfusion with UW solution — Totally 6 L of cold UW solution were infused (aortic: portal =1:1)
  Arms: sole perfusion

SUMMARY:
The study was designed to investigate whether, compared with conventional sole perfusion with high-viscosity solution of University of Wisconsin (UW), sequential perfusion of liver grafts with low-viscosity and high-viscosity preservation solutions could further decrease the incidence of nonanastomotic biliary strictures (NAS) after liver transplantation.

DETAILED DESCRIPTION:
The exact etiology of nonanastomotic biliary strictures (NAS) with a patent hepatic artery after liver transplantation remains unclear so far. Microangiopathy is strongly suspected to be involved in the etiology, so sufficient flushing of peribiliary plexus (PBP) which directly nourishes the donor biliary tree may be pivotal to prevent NAS with a patent hepatic artery.

Solution of University of Wisconsin (UW solution) is a standard for liver graft flushing, but accused of high viscosity and hyperaggregation effect on erythrocytes by ingredient hydroxyethyl starch as well as initial vasoconstriction by high potassium content, which together constitutes a hindrance to solution penetration and thorough flushing of liver microcirculation including PBP. Several studies have revealed the relationship of high viscosity of UW solution with the development of NAS.

The investigators, therefore, have hypothesized that sequential perfusion with low-viscosity and high-viscosity preservation solutions might improve the patency of PBP in contrast with conventional sole perfusion with high-viscosity UW solution, and as a result, the incidence of NAS with a patent hepatic artery after liver transplantation would be significantly decreased.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* ability to provide written informed consent prior to study entry
* receiving a whole liver graft
* primary transplantation

Exclusion Criteria:

* participant in other clinical trials
* fulminant liver failure as the cause of transplantation
* primary biliary cirrhosis, autoimmune hepatitis or primary sclerosing cholangitis as primary liver disease
* retransplantation
* non-liver organ(s) failure prior to study entry
* donor/recipient ABO-blood-group-incompatibility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2004-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with primary non-function (PNF) for safety assessment of sequential perfusion | 1 week
  PNF is defined as non-life-sustaining function of the graft unexplained by vascular complications or rejection, leading to death or retransplantation within postoperative 7 days.
Number of participants with nonanastomotic biliary strictures with a patent hepatic artery | 5 years
  nonanastomotic biliary strictures secondary to hepatic arterial thrombosis or stenosis will be excluded from calculation.

SECONDARY OUTCOMES:
Number of participants with initial poor function (IPF) | 1 week
  IPF is defined as a delayed function restoration with serum AST level greater than 2,000 U/L and prothrombin time greater than 16 seconds postoperative days 2 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Hai Peng, Prof., Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Moench C, Moench K, Lohse AW, Thies J, Otto G. Prevention of ischemic-type biliary lesions by arterial back-table pressure perfusion. Liver Transpl. 2003 Mar;9(3):285-9. doi: 10.1053/jlts.2003.50015. PMID 12619026
- [Background] Pirenne J, Van Gelder F, Coosemans W, Aerts R, Gunson B, Koshiba T, Fourneau I, Mirza D, Van Steenbergen W, Fevery J, Nevens F, McMaster P. Type of donor aortic preservation solution and not cold ischemia time is a major determinant of biliary strictures after liver transplantation. Liver Transpl. 2001 Jun;7(6):540-5. doi: 10.1053/jlts.2001.24641. PMID 11443584
- [Background] Sanchez-Urdazpal L, Gores GJ, Ward EM, Maus TP, Buckel EG, Steers JL, Wiesner RH, Krom RA. Diagnostic features and clinical outcome of ischemic-type biliary complications after liver transplantation. Hepatology. 1993 Apr;17(4):605-9. doi: 10.1002/hep.1840170413. PMID 8477965